CLINICAL TRIAL: NCT02529059
Title: A Phase IV, Open-label, Multi Centre Pilot Study to Assess Changes in Cerebral Function Parameters in Patients Without Perceived Central Nervous System (CNS) Symptoms When Switched From a Fixed Dose Combination of Tenofovir/Emtricitabine/Efavirenz (Atripla®) to a Fixed Dose Combination of Tenofovir/Emtricitabine/Rilpivirine (Eviplera®)
Brief Title: SSAT058: Atripla to Eviplera Switch in Patients Without Central Nervous System Symptoms
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: St Stephens Aids Trust (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SSAT058
Record Dates: First submitted 2015-05-27; First posted 2015-08-19 (Estimated); Last update posted 2017-09-18 (Actual); Status verified 2017-09

CONDITIONS: HIV
MeSH Terms: interventions — Rilpivirine; Tenofovir; Emtricitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Switch from Atripla to Eviplera (Experimental)
  Interventions: Drug: Eviplera

INTERVENTIONS:
Drug: Eviplera — A single-pill fixed dose combination of tenofovir 245mg, emtricitabine 200mg and rilpivirine 25mg once daily for 24 weeks.
  Other Names: Rilpivirine, tenofovir, emtricitabine

SUMMARY:
This study aims to investigate whether substitution of Efavirenz (EFV) as the Tenofovir/Emtricitabine/Efavirenz (TDF/FTC/EFV) fixed-dose combination (FDC) Atripla, with Rilpivirine as the tenofovir/emtricitabine/rilpivirine (TDF/FTC/RPV) fixed-dose combination (FDC) Eviplera, leads to resolution of covert Central Nervous System (CNS) toxicity associated with EFV, continued virological suppression and immunological reconstitution and whether this is associated with an improvement in quality of life, sleep, anxiety/depression and neurocognitive function; the impact of switch on adherence will also be investigated.

DETAILED DESCRIPTION:
Protocol Summary

Study Title: SSAT 058 - A phase IV, open-label, multi centre pilot study to assess the prevalence of objective neurocognitive abnormality in patients without perceived Central Nervous System (CNS) symptoms on tenofovir/emtricitabine/efavirenz Atripla® and the effect of switching to a fixed dose combination of tenofovir/emtricitabine/rilpivirine (Eviplera®).

Proposed Sponsor: St Stephen's AIDS Trust

Chief Investigator: Dr Mark Nelson

Name of Investigational Product: Eviplera®

Name of Active Ingredients: Rilpivirine, tenofovir, emtricitabine

Name of Non Investigational Medicinal Product : NA

Name of Active Ingredients: NA

Phase of Study: Phase IV

Objectives: The objectives of this study are:

Primary objectives

* To describe prevalence pattern, in patients without self-perceived CNS symptoms related to tenofovir/emtricitabine/efavirenz, of the following parameters assessed at baseline:

  * Objective neurocognitive function testing.
  * Self-reported central nervous system symptoms by questionnaire
  * Reported Sleep quality Secondary objectives
* change in measured neurocognitive parameters from baseline to week 4 and 24
* change in sleep scores from baseline to week 4 and 24
* change in symptoms related to CNS toxicity from baseline over 24 weeks
* change in magnetic resonance imaging (MRI) and spectroscopy of brain between baseline and week 24.
* the rate of maintained virological suppression at <50 copies/ml at each visit over 24 weeks
* changes in fasting lipids from baseline over 24 weeks
* change in reported adherence from baseline and to week 24 in:

  * adherence
  * Quality of life
  * Reported anxiety and depression

Study Design: Multi-centre, open-label, single pilot study of 24 weeks. Study visits will take place at screening, baseline (within 36 days of screening visit), weeks 4, 12 and 24.

Substudy of 10 volunteers - MRI scan at baseline and week 24

Indication: HIV-1-infection

Methodology:

* Neurocognitive function testing measured by computerised tasks.
* CNS symptoms and sleep quality determined by questionnaire.
* Changes in CNS metabolites by 1H-MR spectroscopy imaging.

Planned Sample Size: 40 (across 4 centres)

Summary of Eligibility Criteria: HIV-infected individuals on Atripla with a viral load < 50 copies/mL and a CD4 count > 50 cells/mm3.

Number of Study Centres: 4

Duration of Treatment: 24 weeks

Dose and Route of Administration: A single-pill fixed dose combination of tenofovir 245mg, emtricitabine 200mg and rilpivirine 25mg once daily.

Primary Endpoint: Summary of overall prevalence and categorised descriptions of the following measures will be determined at baseline:

* Neurocognitive function scores calculated as composite scores and individual domains.
* Reported CNS symptoms assessed using questionnaire based on Summary of Product Characteristics (SPC) will be scored for severity and reported as both individual and composite scores.
* Sleep Quality assessed by questionnaire at baseline.

Secondary Endpoint:

* change in measured neurocognitive parameters from baseline to week 4 and 24
* change in sleep scores from baseline to week 4 and 24
* change in symptoms related to CNS toxicity from baseline over 24 weeks
* Change in magnetic resonance imaging and spectroscopy of brain between baseline and week 24.
* the rate of maintained virological suppression at <50 copies/ml at each visit over 24 weeks
* changes in fasting lipids from baseline over 24 weeks
* change in reported adherence from baseline and to week 24 in:

  * adherence
  * Quality of life
  * Reported anxiety and depression

ELIGIBILITY:
Inclusion Criteria:

Patient volunteers who meet all of the following criteria are eligible for this trial:

1. Is male or female aged 18 years or above
2. Has HIV-1 infection documented in their medical notes
3. Has signed the Informed Consent Form voluntarily
4. Is willing to comply with the protocol requirements
5. Has been on Atripla for at least 12 weeks before enrolment
6. Has an undetectable HIV-plasma viral load at screening by local assay (single re-test allowed)
7. Has a CD4 cell count at screening >50 cells/mm3
8. Has an estimated glomerular filtration rate (MDRD) >50 ml/min.
9. Has no significant CNS symptoms which may be attributable to EFV.
10. If female and of childbearing potential, is using effective birth control methods (for example, hormonal contraceptive, condom, abstinence, IUD, as agreed by the investigator) and is willing to continue practising these birth control methods during the trial and for at least 30 days after the end of the trial. Note: Women who are postmenopausal for least 2 years, women with total hysterectomy, and women who have a tubal ligation are considered of non-childbearing potential
11. If a heterosexually active male, he is using effective birth control methods and is willing to continue practising these birth control methods during the trial and until follow-up visit

Exclusion Criteria:

Patients meeting 1 or more of the following criteria cannot be selected:

1. Infected with HIV-2
2. Using any concomitant therapy disallowed as per SPC for the study drugs (e.g proton pump inhibitors )
3. Has acute viral hepatitis including, but not limited to, A, B, or C
4. Has chronic hepatitis B and/or C with AST and/or ALT >5 x ULN Note: Patients can enter trial with chronic HBV if HBV-DNA undetectable at screen (and no detectable result in last 6 months) and with chronic HCV if not expected to require treatment during the trial period.
5. Any investigational drug within 30 days prior to the trial drug administration
6. Has ever received rilpivirine in the past
7. Any clinical evidence of baseline resistance mutations, prior to commencing antiretroviral therapy.
8. Known allergy to lactose monohydrate, sunset yellow aluminium lake (E110), and patients with galactose intolerance, the Lapp lactase deficiency, or glucose-galactose malabsorption
9. Severe hepatic impairment (defined as Child-Pugh-Turcotte (CPT) Score C).
10. If female, she is pregnant or breastfeeding
11. Screening blood result with any grade 3/4 toxicity according to Division of AIDS (DAIDS) grading scale, except: asymptomatic grade 3 glucose, amylase or lipid elevation or asymptomatic grade 4 triglyceride elevation (re-test allowed).
12. Any condition (including drug/alcohol abuse) or laboratory results which, in the investigator's opinion, interfere with assessments or completion of the trial.
13. If participating in the MR Imaging substudy, any contraindications to magnetic resonance scanning according to local radiology guidelines (to be assessed by MR Spectroscopy Imaging Department)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-11; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Change in neuropsychiatric and central nervous system (CNS) parameters after switching from Atripla to TDF/FTC/RPV at 4 weeks compared to baseline, as measured by the proportion of patients experiencing grade 2-4 neuropsychiatric and CNS toxicity | 4 Weeks compared to baseline
  As defined by the ACTG Adverse event scale and collected by CNS questionnaire.
Change in neuropsychiatric and central nervous system (CNS) parameters after switching from Atripla to TDF/FTC/RPV at 4 weeks compared to baseline, as measured by the median number of grade 2-4 neuropsychiatric and CNS toxicity | 4 Weeks compared to baseline
  As defined by the ACTG adverse event scale and collected by CNS questionnaire.
Change in neuropsychiatric and central nervous system (CNS) parameters after switching from Atripla to TDF/FTC/RPV at 4 weeks compared to baseline, as measured by the median CNS score. | 4 Weeks compared to baseline
  Derived from the sum of toxicity of all grades collected in the CNS questionnaire.
Change in neuropsychiatric and central nervous system (CNS) parameters after switching from Atripla to TDF/FTC/RPV at 4 weeks compared to baseline, as measured by the change in sleep score using the Pittsburgh Sleep Questionnaire. | 4 Weeks compared to baseline

SECONDARY OUTCOMES:
Change in neuropsychiatric and central nervous system (CNS) parameters after switching from Atripla to TDF/FTC/RPV at 12 & 24 weeks compared to baseline, as measured by proportion of patients experiencing grade 2-4 neuropsychiatric and CNS toxicity. | 12 and 24 weeks compared to baseline
  As defined by the ACTG adverse event scale and collected by CNS questionnaire.
Change in neuropsychiatric and central nervous system (CNS) parameters after switching from Atripla to TDF/FTC/RPV at 12 and 24 weeks compared to baseline, as measured by the median number of grade 2-4 neuropsychiatric and CNS toxicity. | 12 and 24 weeks compared to baseline
  As defined by the ACTG adverse event scale and collected by CNS questionnaire.
Change in neuropsychiatric and central nervous system (CNS) parameters after switching from Atripla to TDF/FTC/RPV at 12 and 24 weeks compared to baseline, as measured by the median CNS score | 12 and 24 weeks compared to baseline
  Median CNS score is derived from the sum of toxicity of all grades collected in the CNS questionnaire.
Change in neuropsychiatric and central nervous system (CNS) parameters after switching from Atripla to TDF/FTC/RPV at 12 and 24 weeks compared to baseline, as measured by change in sleep score using the Pittsburgh Sleep Questionnaire. | 12 and 24 weeks compared to baseline
Change in neuropsychiatric and CNS parameters as measured by the change in the Hospital Anxiety and Depression Scale (HADS) at 4, 12 and 24 weeks as compared with baseline. | 4, 12 and 24 weeks compared to baseline
Proportion of patients with undetectable viral load (by local assay) at weeks 4, 12 and 24. | 4, 12 and 24 weeks compared to baseline
Proportion of patients with viral load below 400 copies/mL at weeks 4, 12 and 24. | 4, 12 and 24 weeks compared to baseline
Change in CD4+ count at week 12 and 24 compared to baseline. | 12 and 24 weeks compared to baseline
Proportion of patients with grade 2-4 laboratory adverse events (excluding lipids) and proportion of patients with grade 2-4 non-CNS adverse events at 4, 12 and 24 weeks compared with baseline. | 4, 12 and 24 weeks compared to baseline
Change in mean fasting cholesterol (total, HDL, LDL and total:HDL ratio) and triglycerides after 4, 12 and 24 weeks compared with baseline. | 4, 12 and 24 weeks compared to baseline
Change in quality of life (as assessed by EQ-5D questionnaire) at 4, 12 and 24 weeks compared with baseline. | 4, 12 and 24 weeks compared to baseline
Change in neurocognitive function as determined by computerised neurocognitive assessment (no computerised cognitive testing at week 12) | 4, 12 and 24 weeks compared to baseline
Change in neurocognitive function as determined by Instrumental Activities of Daily Life (IADL) questionnaire | 4, 12 and 24 weeks compared to baseline
Change in adherence as measured by the adherence questionnaire: Medication Adherence Self-Report Inventory (M-MASRI) at 12 and 24 weeks compared with baseline. | 12 and 24 weeks compared to baseline
Change in cerebral MR-measurable imaging modalities at 24 weeks compared with baseline. | 24 weeks compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Mark Nelson, Principal Investigator — St Stephen's AIDs Trust
Locations (3):
- United Kingdom (3):
  - Brighton & Sussex University Hospitals Nhs Trust, Brighton
  - St. Mary's Hospital, London
  - St. Stephen's Centre, London